CLINICAL TRIAL: NCT05198622
Title: Can Chronic Post-surgical Pain be Reduced by Preserving Intercostobrachial Nerve During Axillary Lymph Node Dissection? : A Randomized Controlled Trial
Acronym: PAINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Ibtissam Bin Khalid, Principal Investigator, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-21-28
Record Dates: First submitted 2022-01-09; First posted 2022-01-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Chronic Pain; Intercostobrachial Nerve Injury
Keywords: Chronic Pain; Breast Surgery; Breast Cancer; Intercostobrachial Nerve Injury
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostobrachial Nerve Preservation Arm (Experimental): Intercostobrachial nerve preserving axillary lymph node dissection will be carried out. Post-operatively, the patients will be monitored in the post anesthesia care unit (PACU). Acute Post-Operative pain will be controlled using a standardized pain management regimen in accordance with World Health Organization (WHO) analgesia ladder. The patients will be discharged from PACU and admitted to surgical ward once numerical rating score (NRI) is below 4.
  Interventions: Procedure: Intercostobrachial Nerve Preserving Axillary Lymph Node Dissection
- Intercostobracial Nerve Sacrifice Arm (Active Comparator): Intercostobrachial nerve sacrificing axillary lymph node dissection will be carried out. Post-operatively, the patients will be monitored in the post anesthesia care unit (PACU). Acute Post-Operative pain will be controlled using a standardized pain management regimen in accordance with World Health Organization (WHO) analgesia ladder. The patients will be discharged from PACU and admitted to surgical ward once numerical rating score (NRI) is below 4.
  Interventions: Procedure: Intercostobrachial Nerve Sacrificing Axillary Lymph Node Dissection

INTERVENTIONS:
Procedure: Intercostobrachial Nerve Preserving Axillary Lymph Node Dissection — A single standardized technique will be used in all of the patients. For patients undergoing mastectomy, ALND will be carried out using the incision given for mastectomy. A separate incision may be required for patients undergoing breast conservation surgery. Flaps of skin and subcutaneous tissue will be raised and dissection will be carried out till the edge of pectoralis major muscle. Clavipectoral fascia will be opened to gain access to axillary fat and the nodes. These will be removed en block and the intercostobrachial nerve will be completely preserved during this dissection.
  All of the surgeons carrying out the intervention would have completed formal training (Fellowship Level) in breast surgery.
  Arms: Intercostobrachial Nerve Preservation Arm
Procedure: Intercostobrachial Nerve Sacrificing Axillary Lymph Node Dissection — A single standardized technique will be used in all of the patients. For patients undergoing mastectomy, ALND will be carried out using the incision given for mastectomy. A separate incision may be required for patients undergoing breast conservation surgery. Flaps of skin and subcutaneous tissue will be raised and dissection will be carried out till the edge of pectoralis major muscle. Clavipectoral fascia will be opened to gain access to axillary fat and the nodes. These will be removed en block and the intercostobrachial nerve will be sacrificed during this dissection.
  All of the surgeons carrying out the intervention would have completed formal training (Fellowship Level) in breast surgery.
  Arms: Intercostobracial Nerve Sacrifice Arm

SUMMARY:
Intercostobrachial nerve (ICBN) is a cutaneous nerve that provides sensation to the lateral chest, upper medial arm and axilla. It arises from the second intercostal nerve and leave intercostal space at the level of midaxillary line. It then pierces the serratus anterior muscle and enters axilla. Intercostobrachial nerve is encountered during axillary lymph node dissection (ALND) while mobilizing axillary contents laterally off the chest wall and tends to tether axillary contents to the lateral chest wall. Many surgeons routinely sacrifice it as doing so makes mobilization easier and allow exposure of long thoracic neve. Currently there is no consensus on the usefulness of preserving intercostobrachial nerve.

According to a 2020 systemic review and meta-analysis, prevalence of CPSP/ PPSP following breast cancer surgery ranged from 2% to 78% and pooled prevalence was found to be 35%. Higher prevalence was associated with ALND. Several risk factors have been identified which contribute to the development of PPSP. These include; Preexisting pain, preoperative opioid exposure, genetics, psychological factors such as anxiety, depression or catastrophizing, intensity of acute postoperative pain and nerve injury during surgery.

As a result of nerve injury, damaged and non-damaged nerve fibers start generating action potential spontaneously. These are considered ectopic inputs as they do not arise from peripheral terminals. These inputs lead to the development of central sensitization, which is a state of exaggerated functional response of neurons involved in the pain pathway. This increased sensitization results due to increased membrane excitability, enhanced synaptic efficacy and decreased inhibition.

The aim of the present trial is to investigate the effect of ICBN preservation on chronic/ persistent post surgical pain (CPSP/ PPSP). This will be achieved through a randomized control trial with CPSP/ PPSP as a primary outcome measure. Secondary outcome measures will include Health Related Quality of Life (HRQoL), operating time, lymph node yield, functional status of ipsilateral shoulder, post-operative complications and post-operative use of opioid analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above.
* Known cases of invasive breast Cancer.
* Undergoing Axillary Lymph Node Dissection (ALND) alone, ALND with mastectomy or ALND with breast conservation surgery (BCS)
* Capacity to give informed consent

Exclusion Criteria:

* Chronic diseases limiting motion of shoulder such as neuropathies, history of trauma and autoimmune diseases.
* Patients undergoing redo axillary lymph node dissection.
* Patients undergoing bilateral axillary lymph node dissection.
* History of chronic pain lasting more than 3 months. Potential causes include: arthritis, backache, fibromyalgia, Irritable bowel disease, irritable bowel syndrome and different types of headache.
* M1 stage of the TNM staging system at the time of initial diagnosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Persistent Post-Surgical Pain (PPSP) using Brief Pain Inventory-Short Form (BPI SF) | Baseline (Pre-Operatively)
  BPI SF is a validated tool for the measurement of chronic pain. It assesses average pain intensity over the past 24 hour period. It defines pain as follows:
  Mild Pain: Score 1-4 Moderate Pain: Score 5-6 Severe Pain: Score 7-10 Recall Period: Last 24 hours
Persistent Post-Surgical Pain (PPSP) using Brief Pain Inventory-Short Form (BPI SF) | 2 Weeks (Post-Operatively)
  BPI SF is a validated tool for the measurement of chronic pain. It assesses average pain intensity over the past 24 hour period. It defines pain as follows:
  Mild Pain: Score 1-4 Moderate Pain: Score 5-6 Severe Pain: Score 7-10 Recall Period: Last 24 hours
Persistent Post-Surgical Pain (PPSP) using Brief Pain Inventory-Short Form (BPI SF) | 3 Months (Post-Operatively)
  BPI SF is a validated tool for the measurement of chronic pain. It assesses average pain intensity over the past 24 hour period. It defines pain as follows:
  Mild Pain: Score 1-4 Moderate Pain: Score 5-6 Severe Pain: Score 7-10 Recall Period: Last 24 hours
Persistent Post-Surgical Pain (PPSP) using Brief Pain Inventory-Short Form (BPI SF) | 6 Months (Post-Operatively)
  BPI SF is a validated tool for the measurement of chronic pain. It assesses average pain intensity over the past 24 hour period. It defines pain as follows:
  Mild Pain: Score 1-4 Moderate Pain: Score 5-6 Severe Pain: Score 7-10 Recall Period: Last 24 hours

SECONDARY OUTCOMES:
Health Related Quality of Life using Functional Assessment of cancer therapy-Breast form (FACT-B) | Baseline (Pre-Operatively), 2 weeks (Post-Operatively), 3 months (Post-Operatively) and 6 months (Post-Operatively)
  FACT-B is a 37 item, validated tool for the measurement of health of health related quality of life (HRQoL). It consists of five subscales: Physical well being, emotional well being, social well being, functional well being and a breast cancer-specific subscale. Items are rated from 0 (not at all) to 4 (very much) and a total score is calculated. The total score ranges from 0-148. Lower score indicates a better health related quality of life.
  Recall Period: Last 7 Days
Functional Status of Ipsilateral Shoulder using Shoulder Pain and Disability Index (SPADI) Questionnaire | Baseline (Pre-Operatively), 2 weeks (Post-Operatively), 3 months (Post-Operatively) and 6 months (Post-Operatively)
  SPADI is a validated tool for the measurement of shoulder pain and disability. It is composed of pain component and functional assessment component. Each item in score component is rated from 0 (no pain) to 10 (worst imaginable pain) whereas items in functional assessment component are rated from 0 (no difficulty) to 10 (so difficult it requires help). The total score is expressed as a percentage. A higher score indicates more disability.
  Recall Period: Last 7 Days
Operating Time (Minutes) | Intraoperative
  Operating Time is the time duration from incision to the closure. It will be measured in minutes.
Lymph Node Yield | Intraoperative
  Lymph node yield is the total number of benign or malignant lymph nodes found in the axillary lymph node dissection specimen at the time of histopathological analysis.
Post-Operative Complications as per Clavien Dindo Classification (CDC) | From the time of intervention to 30 days (Post-Operatively)
  Clavien Dindo Classification divides the severity of post-operative complications based on the level of medical intervention needed. CDC is as following:
  Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgesics, diuretics, electrolytes and physiotherapy. This Grade also includes wound infections opened at the bedside.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for Grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III (a): intervention not under general anesthesia Grade III (b): intervention under general anesthesia Grade IV: Life-threatening complication (including complications of the Central Nervous System) requiring Intermediate Care/Intensive Care Unit management Grade V: Death of a patient
Post-Operative usage of Opioid Analgesics | 2 weeks (Post-Operatively), 3 months (Post-Operatively) and 6 months (Post-Operatively)
  Type of opioid analgesic and prescribed daily dose in the post-operative period
Adverse Events | From the time of intervention to 6 months (Post-Operatively)
  All adverse events will be documented on case report forms. The data management committee (DMC) will review these adverse events and determine if these are due to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ibtissam Bin Khalid, MBBS, Principal Investigator — Shaukat Khanum Memorial Cancer Hospital & Research Center
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital & Research Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Cohen JC, Devasenapathy N, Hong BY, Kheyson S, Lu D, Oparin Y, Kennedy SA, Romerosa B, Arora N, Kwon HY, Jackson K, Prasad M, Jayasekera D, Li A, Guarna G, Natalwalla S, Couban RJ, Reid S, Khan JS, McGillion M, Busse JW. Prevalence and intensity of persistent post-surgical pain following breast cancer surgery: a systematic review and meta-analysis of observational studies. Br J Anaesth. 2020 Sep;125(3):346-357. doi: 10.1016/j.bja.2020.04.088. Epub 2020 Jun 28. PMID 32611524
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Abdullah TI, Iddon J, Barr L, Baildam AD, Bundred NJ. Prospective randomized controlled trial of preservation of the intercostobrachial nerve during axillary node clearance for breast cancer. Br J Surg. 1998 Oct;85(10):1443-5. doi: 10.1046/j.1365-2168.1998.00843.x. PMID 9782034
- [Background] Torresan RZ, Cabello C, Conde DM, Brenelli HB. Impact of the preservation of the intercostobrachial nerve in axillary lymphadenectomy due to breast cancer. Breast J. 2003 Sep-Oct;9(5):389-92. doi: 10.1046/j.1524-4741.2003.09505.x. PMID 12968959
- [Background] Salmon RJ, Ansquer Y, Asselain B. Preservation versus section of intercostal-brachial nerve (IBN) in axillary dissection for breast cancer--a prospective randomized trial. Eur J Surg Oncol. 1998 Jun;24(3):158-61. doi: 10.1016/s0748-7983(98)92793-7. PMID 9630850
- [Background] Kaur N, Kumar R, Jain A, Saxena AK. Sensory Changes and Postmastectomy Pain Following Preservation of Intercostobrachial Nerve in Breast Cancer Surgery: a Prospective Randomized Study. Indian J Surg Oncol. 2021 Mar;12(1):108-113. doi: 10.1007/s13193-020-01193-5. Epub 2020 Sep 5. PMID 33814840
- [Background] Taira N, Shimozuma K, Ohsumi S, Kuroi K, Shiroiwa T, Watanabe T, Saito M. Impact of preservation of the intercostobrachial nerve during axillary dissection on sensory change and health-related quality of life 2 years after breast cancer surgery. Breast Cancer. 2014 Mar;21(2):183-90. doi: 10.1007/s12282-012-0374-x. Epub 2012 Aug 30. PMID 22932759
- [Background] Chirappapha P, Arunnart M, Lertsithichai P, Supsamutchai C, Sukarayothin T, Leesombatpaiboon M. Evaluation the effect of preserving intercostobrachial nerve in axillary dissection for breast cancer patient. Gland Surg. 2019 Dec;8(6):599-608. doi: 10.21037/gs.2019.10.06. PMID 32042666
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536